CLINICAL TRIAL: NCT02360410
Title: Promoting Adolescent Health Through Personalized Feedback
Brief Title: Check Yourself Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laura Richardson (Other)
Responsible Party: Sponsor-Investigator, Laura Richardson, Professor of Pediatrics, University of Washington and Investigator, Seattle Children's Research Institute, Seattle Children's Hospital
Organization: Seattle Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 6 R40MC26817-01-01
Record Dates: First submitted 2015-02-05; First posted 2015-02-10 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Health Risk Behaviors; Health Care Services Quality of Care
MeSH Terms: conditions — Health Risk Behaviors

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Check Yourself App With Feedback (Experimental): Adolescents complete Check Yourself, an electronic health screening app and receive personalized, motivational feedback on their health behaviors prior to their primary care appointment. Key components of Check Yourself include the provision of age normative feedback, goal setting strategies, and strategies to highlight discrepancies. Primary care providers receive a summary report of health risk behaviors from Check Yourself prior to their adolescent patient's primary care appointment.
  Interventions: Behavioral: Check Yourself App with Feedback
- Usual Care (No Intervention): Participants are asked to complete health risk screening on a tablet computer. No personalized feedback is provided to adolescents and primary care providers do not receive a summary report of the adolescent's health risk behaviors.

INTERVENTIONS:
Behavioral: Check Yourself App with Feedback
  Arms: Check Yourself App With Feedback

SUMMARY:
The proposed study is a randomized controlled trial that compares the effectiveness of an electronic personalized health screening app incorporating motivational feedback (i.e., "Check Yourself") to usual care. The purpose of this study is to determine whether Check Yourself is more effective than usual care in reducing health risk behaviors and improving quality of care among adolescents receiving primary health care services.

ELIGIBILITY:
Inclusion Criteria:

* Eligible individuals will be 13-18 years old who have an appointment to see a provider at a participating clinic and will be able to read and comprehend English.

Exclusion Criteria:

* Individuals will be excluded from the study if:

  * they do not meet age requirements,
  * do not have an appointment at a participating clinic,
  * lack the means to complete follow-up interviews (i.e., has neither telephone not internet access),
  * have a sibling who has/is being enrolled in the study and/or
  * are not able to read or comprehend English.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 300 (Actual)
Dates: Start 2015-02; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Number of Health risk behaviors | 3 months
  Total count health-risk behaviors at 3-month follow-up (Score range= 0-13) adjusted by total number of baseline risk behaviors (with risk cut-off): ≥2 sugar-sweetened beverages consumed/day; ≤3 servings fruits/vegetables consumed/day; ≤3 days with 60+ minutes exercise during typical week; ≥3 hours of screen time during typical school day; ≤7 hours of sleep during typical night; not "always" using seatbelt; not "always" using helmet when bicycling; having driven under the influence of substances; days of alcohol consumption in last 30 days (risk based on age: ≥1 day/30 days (ages 13-15), ≥2 days/30 days (ages 16-17), or ≥3 days/30 days (age 18)) and/or number of drinks/drinking episode (risk based on age and sex: ≥3 (Girls 13-17; Boys 13), ≥4 (Girls 18; Boys 14-15), or ≥5 (Boys 16-18)); any tobacco use; any marijuana/other drugs use; not using birth control during last sexual intercourse and/or not "always" using a condom; and ≥10 score on PHQ-9.
Number of risk behaviors counseled on during primary care appointment | 1 day
  Number of adolescent-reported high risk health risk behaviors discussed with the healthcare provider during the primary care visit (Score range: 0-13) adjusted for the total number of health risk behaviors reported at baseline. Receipt of counseling/discussion assessed using an adapted version of the Adolescent Report of the Visit (AROV). The AROV includes counseling on the following behaviors: 1) sweetened beverage consumption; 2) fruit/vegetable consumption; 3) physical activity amount; 4) screen time (i.e., watching TV, playing video games, surfing the web, or texting); 5) sleep duration; 6) seat belt use; 7) helmet use while bicycling; 8) drinking/using drugs while driving; 9) alcohol use; 10) tobacco use; 11) marijuana and/or other drug use; 12) condom and/or birth control use; 13) depression and moods.

SECONDARY OUTCOMES:
Adolescent Satisfaction with Care | 1 day
  Adolescent satisfaction with care will be assessed using the total score on the 8-item Client Satisfaction Questionnaire (CSQ-8) at 1-day follow-up.
Interval Receipt of Care | 3 months
  Dichotomous variable indicating receipt of any follow-up care to address risk behaviors identified at baseline adjusted for baseline number of health risk behaviors.
Motivation for Health Behavior Change | 1 day
  Assessment of adolescent reported motivation to change overall health using a Readiness to Change Ruler.
Specific Health Risk Behavior Change | 3 months
  Reported level for each specific health risk behavior at 3 months adjusting for baseline level of that specific behavior. Specific individual behaviors include: A.) number of: sweetened beverages consumed in a typical day; fruits and vegetables consumed in a typical day; days with >60 minutes of physical activity in an average week; hours of screen time on a typical day; hours of sleep on a typical night; days in which alcohol was consumed in the prior month; alcoholic drinks typically consumed per occasion; any tobacco use in the prior month (yes/no); days using marijuana in the past month; B) Score on the nine item Patient Health Questionnaire (27 point scale); C) Frequency of: seatbelt use in a car (4-point scale); helmet use while bicycling (4-point scale); condom use with sexual intercourse (4-point scale); D) Use of any form of birth control at last sexual intercourse (yes/no); and E) Driving under the influence of a substance (yes/no).

OTHER OUTCOMES:
Adolescent Perceived Support from their Primary Care Provider | 1 day
  The total score on the Health Care Climate Questionnaire (HCCQ),) will be used to assess adolescent self-report of perceived autonomy support from their primary care provider.
Adolescent Health Self-Efficacy | 1 day
  The total score on the Health Self Efficacy Scale will be used to assess adolescent self-report of perceived confidence in ability to execute health behaviors.

CONTACTS AND LOCATIONS:
Overall Officials: Laura P Richardson, MD MPH, Principal Investigator — Seattle Children's Hospital
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States

REFERENCES:
- [Derived] Richardson LP, Zhou C, Gersh E, Spielvogle H, Taylor JA, McCarty CA. Effect of Electronic Screening With Personalized Feedback on Adolescent Health Risk Behaviors in a Primary Care Setting: A Randomized Clinical Trial. JAMA Netw Open. 2019 May 3;2(5):e193581. doi: 10.1001/jamanetworkopen.2019.3581. PMID 31074815